CLINICAL TRIAL: NCT03113396
Title: A Double-blind, Placebo-controlled, Cross-over Study Using Baclofen in the Treatment of Rumination Syndrome
Brief Title: Baclofen for Rumination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S53446
Record Dates: First submitted 2017-03-21; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Rumination; Supra-gastric Belching
MeSH Terms: conditions — Rumination Syndrome | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- baclofen (Experimental): Patients will receive baclofen (10mg t.i.d) for 2 weeks, thereafter they will be crossed over to the alternative treatment, which is placebo (identically looking capsules). After 2 weeks of treatment, patients will undergo a High Resolution Impedance Manometry (HRiM) measurement, with meal. We will record for in total 2 hours. Patients are asked to fill out questionnaires concerning their overall wellbeing.
  Interventions: Drug: Baclofen
- placebo (Placebo Comparator): Patients will receive placebo for 2 weeks, thereafter they will be crossed over to the alternative treatment, which is baclofen (10mg t.i.d) (identically looking capsules). After 2 weeks of treatment, patients will undergo a High Resolution Impedance Manometry (HRiM) measurement, with meal. We will record for in total 2 hours. Patients are asked to fill out questionnaires concerning their overall wellbeing.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Baclofen — baclofen oral, 10mg, tid for 2 weeks (or placebo, identically looking capsules) after 2 weeks, patients undergo a High Resolution Impedance Manometry measurement with a meal period. Patients will fill out questionnaires concerning overall wellbeing.
  Other Names: Lioresal
  Arms: baclofen
Drug: Placebo oral capsule — placebo oral, tid for 2 weeks after 2 weeks, patients undergo a High Resolution Impedance Manometry measurement with a meal period. Patients will fill out questionnaires concerning overall wellbeing.
  Arms: placebo

SUMMARY:
Patients with a clinical suspicion of rumination syndrome and/or supra-gastric belching are randomized into baclofen or placebo for 2 weeks (10mg, tid). thereafter, they undergo a high resolution impedance manometry measurement, were they receive a solid meal, and recordings continue for another hour. Thereafter, they will receive the alternative treatment, after which they will undergo a second high resolution impedance manometry measurement. Patients are asked to fill out questionnaires during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of rumination syndrome and/or supra-gastric belching.
* Sexually active women of child bearing potential participating in the study must use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception.
* 18 to 75 years old.
* Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

* Systemic diseases, known to affect esophageal motility.
* Surgery in thorax or in the upper part of the abdomen.
* Treatment with baclofen prior to the start of the study.
* Significant neurological, respiratory, hepatic, renal, haematological, cardiovascular, metabolic or gastrointestinal cerebrovascular disease as judged by the investigator.
* Pregnancy or breast feeding.
* History of poor compliance. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent. (well-controlled depression is allowed).
* History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Overall wellbeing of the patients, assessed by an overall treatment evaluation questionnaire. | 2 weeks treatment
  patients fill out questionnaires concerning overall wellbeing, during the 2 weeks of treatment. Results of these questionnaires will be compared between both conditions (baclofen and placebo).

SECONDARY OUTCOMES:
objective measurement of rumination / supra-gastric belching, using high resolution impedance manometry monitoring | 2 weeks treatment
  High Resolution impedance Manometry monitoring will be performed, with a meal. We will look at the number of times patients push an event marker, the number of time patients ruminate or have supra-gastric belching or have reflux episodes, or have transient lower esophageal sphincter relaxations, both before and after the meal. And we will compare these outcomes between placebo and baclofen.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pauwels A, Broers C, Van Houtte B, Rommel N, Vanuytsel T, Tack J. A Randomized Double-Blind, Placebo-Controlled, Cross-Over Study Using Baclofen in the Treatment of Rumination Syndrome. Am J Gastroenterol. 2018 Jan;113(1):97-104. doi: 10.1038/ajg.2017.441. Epub 2017 Dec 5. PMID 29206813